CLINICAL TRIAL: NCT01180933
Title: Dietary Supply of Docosahexaenoic Acid (DHA) and 5-methyl-tetrahydro-folate (MTHF) During the Second Half of Pregnancy and Early Infancy
Brief Title: Fish Oil and Folate Supplementation During Pregnancy
Acronym: NUHEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: European Union (Other)
Responsible Party: Prof. Dr. Berthold Koletzko, Ludwig-Maximilians University of Munich
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01111
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-06

CONDITIONS: Perinatal DHA and Folate Status; Neurological Development
Keywords: docosahexaenoic acid; folate; neurological development; allergies; long term consequences for the offspring; allergy risk
MeSH Terms: conditions — Hypersensitivity | interventions — Fish Oils; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- fish oil (Experimental): the participating women receive a milk based supplement providing vitamins and mineral as recommended for pregnant women and 500 mg DHA and 150 eicosapentaenoic acid per day from gestational week 22 until delivery
  Interventions: Dietary Supplement: fish oil
- folate (Experimental): the participating women receive a milk based supplement providing vitamins and mineral as recommended for pregnant women and 400 µg folate (methyltetrahydrofolate)per day from gestational week 22 until delivery
  Interventions: Dietary Supplement: folate
- fish oil + folate (Experimental): the participating women receive a milk based supplement providing vitamins and mineral as recommended for pregnant women and 500 mg DHA, 150 mg eicosapentaenoic acid and 400 µg MTHF per day from gestational week 22 until delivery
  Interventions: Dietary Supplement: fish oil + folate
- placebo (Placebo Comparator): the participating women receive a milk based supplement providing vitamins and mineral as recommended for pregnant women from gestational week 22 until delivery
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: fish oil — 400 mg of DHA and 150 mg of eicosapentaenoic acid per day
  Arms: fish oil
Dietary Supplement: folate — 400 µg per day
  Arms: folate
Dietary Supplement: fish oil + folate — 500 mg DHA, 150 mg eicosapentaenoic acid, 400 µg MTHF per day
  Arms: fish oil + folate
Dietary Supplement: placebo — only vitamins and minerals as recommended, but no fish oil or folate
  Arms: placebo

SUMMARY:
Pregnant women are randomised to supplementation with fish oil, methyl tetrahydro folic acid, both or a placebo during the second half of pregnancy. Biochemical measures are determined in maternal blood during pregnancy and in cord blood.

Non invasive follow up examinations of infants at ages 4, 5.5, 6.5, 7.5, 8, 9 and 9.5 years focus on long term effects of supplementation anthropometric development, neurological development and allergy risk.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* gestation <20 week at enrollment
* intention to deliver in one of the study centers
* body weight at time of enrollment from 50 kg to 92 kg

Exclusion Criteria:

* serious chronic illness (eg, diabetes, hepatitis)
* use fish oil supplements since the beginning of pregnancy
* use of folate or vitamin B-12 supplements after gestation week 16

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 315 (Actual)
Dates: Start 2001-11; Primary Completion 2003-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
percentage contribution of docosahexaenoic acid (DHA) to total phospholipid fatty acids in cord blood | labour
  the biochemical efficacy of supplementation during pregnancy is tested by measuring the DHA content of cord blood phospholipids, as direct supplementation (fish oil) or increased perfusion of the placenta (MTHF) could both influence this parameter

SECONDARY OUTCOMES:
neurological and cognitive development of the offspring | age 4 years, 5.5 years, 6.5 years, 7.5 years, 8 years, 9 years, 9.5 years
  non invasive, age adequate, tests of neurological and cognitive function are performed at various ages of the offspring
weight development | age 4 years, 5.5 years, 6.5 years, 8 years, 9.5 years
  body weight (including weight of fat and non fat mass by bioelectrical impedance at later ages) is determined
height | age 4 years, 5.5 years, 6.5 years, 8 years, 9.5 years
  body height is measured at ages 4 years, 5.5 years, 6.5 years, 8 years, 9.5 years
life style and diet | age 4 years, 5.5 years, 6.5 years, 7.5 years, 8 years, 9 years, 9.5 years
  information on medical history, life sytyle and dietary habits is collected via questionnaires and non invasivly collected of biological samples (urine, cheek cells)
electroencephalography (EEG) | age 8 years and 9.5 years
  at age 8 years and 9.5 years an EEG is obtained while the children are performing defined tests

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Prof., Study Director — Dr. von Hauner Childrens Hospital, Ludwig-Maximilians-University Munich
Locations (3):
- Dr. von Hauner Childrens Hospital, Ludwig-Maximilians-University, Munich, Germany
- University of Pecs, Pécs, Hungary
- Department of Paediatrics, University of Granada, Granada, Spain

REFERENCES:
- [Result] Krauss-Etschmann S, Shadid R, Campoy C, Hoster E, Demmelmair H, Jimenez M, Gil A, Rivero M, Veszpremi B, Decsi T, Koletzko BV; Nutrition and Health Lifestyle (NUHEAL) Study Group. Effects of fish-oil and folate supplementation of pregnant women on maternal and fetal plasma concentrations of docosahexaenoic acid and eicosapentaenoic acid: a European randomized multicenter trial. Am J Clin Nutr. 2007 May;85(5):1392-400. doi: 10.1093/ajcn/85.5.1392. PMID 17490978
- [Derived] Catena A, Munoz-Machicao JA, Torres-Espinola FJ, Martinez-Zaldivar C, Diaz-Piedra C, Gil A, Haile G, Gyorei E, Molloy AM, Decsi T, Koletzko B, Campoy C. Folate and long-chain polyunsaturated fatty acid supplementation during pregnancy has long-term effects on the attention system of 8.5-y-old offspring: a randomized controlled trial. Am J Clin Nutr. 2016 Jan;103(1):115-27. doi: 10.3945/ajcn.115.109108. Epub 2015 Nov 11. PMID 26561619
- [Derived] Campoy C, Escolano-Margarit MV, Ramos R, Parrilla-Roure M, Csabi G, Beyer J, Ramirez-Tortosa MC, Molloy AM, Decsi T, Koletzko BV. Effects of prenatal fish-oil and 5-methyltetrahydrofolate supplementation on cognitive development of children at 6.5 y of age. Am J Clin Nutr. 2011 Dec;94(6 Suppl):1880S-1888S. doi: 10.3945/ajcn.110.001107. Epub 2011 Aug 17. PMID 21849596
- [Derived] Escolano-Margarit MV, Ramos R, Beyer J, Csabi G, Parrilla-Roure M, Cruz F, Perez-Garcia M, Hadders-Algra M, Gil A, Decsi T, Koletzko BV, Campoy C. Prenatal DHA status and neurological outcome in children at age 5.5 years are positively associated. J Nutr. 2011 Jun;141(6):1216-23. doi: 10.3945/jn.110.129635. Epub 2011 Apr 27. PMID 21525247